CLINICAL TRIAL: NCT02192970
Title: Bevacizumab Against Recurrent Retinal Detachment
Acronym: BEARRD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2014-0931; A536070 (Other: UW Madison); SMPH/OPHTHAL&VIS SCI (Other: UW Madison)
Record Dates: First submitted 2014-07-15; First posted 2014-07-17 (Estimated); Results first posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Retinal Detachment; Proliferative Vitreoretinopathy
Keywords: Retinal detachment; Proliferative vitreoretinopathy
MeSH Terms: conditions — Retinal Detachment; Vitreoretinopathy, Proliferative | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bevacizumab (Experimental): Pars plana vitrectomy will be performed in the typical manner. After laser retinopexy and prior to air-gas exchange, intravitreal bevacizumab will be administered through the trocar. Either perfluoropropane (C3F8) or sulfur hexafluoride (SF6) gas will then be administered for long-term retinal tamponade and the vitrectomy ports closed in the usual manner.
  Interventions: Drug: Bevacizumab
- Chart review (No Intervention): Review records over the past 5 years of patients who underwent vitrectomy for retinal detachment repair to found out the percentage of those who had re-detachment of the retina within 6 months after surgery.

INTERVENTIONS:
Drug: Bevacizumab
  Other Names: Avastin
  Arms: Bevacizumab

SUMMARY:
The investigators hypothesize that bevacizumab instilled into the vitreous after primary retinal detachment surgery will reduce the formation of proliferative vitreoretinopathy and subsequent retinal re-detachment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Eyes with rhegmatogenous retinal detachment

Exclusion Criteria:

* Presence of PVR
* Need for a procedure other than primary PPV such as a scleral buckle with or without PPV, laser retinopexy, or pneumatic retinopexy.
* Recent intravitreal injection of an anti-VEGF agent less than 3 months prior
* Secondary retinal detachment repair
* Use of silicone oil as tamponade agent
* Patients less than 18 years of age
* Pregnancy
* Known allergy or contraindication to intravitreal bevacizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2015-01-21 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Altaweel, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- [Background] Pennock S, Kim D, Mukai S, Kuhnle M, Chun DW, Matsubara J, Cui J, Ma P, Maberley D, Samad A, Van Geest RJ, Oberstein SL, Schlingemann RO, Kazlauskas A. Ranibizumab is a potential prophylaxis for proliferative vitreoretinopathy, a nonangiogenic blinding disease. Am J Pathol. 2013 May;182(5):1659-70. doi: 10.1016/j.ajpath.2013.01.052. Epub 2013 Apr 9. PMID 23582767
- See also: Related Info — http://pubmed.gov

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The comparison arm is a chart review, participants were not enrolled in prospective study.
Groups:
- Bevacizumab: Pars plana vitrectomy will be performed in the typical manner. After laser retinopexy and prior to air-gas exchange, intravitreal bevacizumab will be administered through the trocar. Either perfluoropropane (C3F8) or sulfur hexafluoride (SF6) gas will then be administered for long-term retinal tamponade and the vitrectomy ports closed in the usual manner.
  Bevacizumab
Period: Overall Study
Arm/Group | Bevacizumab | Chart Review
Started | 101 | 195
Completed | 95 | 195
Not Completed | 6 | 0
Not completed — Lost to Follow-up | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab | Chart Review | Total
Number analyzed (Participants) | 101 | 195 | 296
Age, Continuous [Mean (Full Range); unit: years] | 61.4 [24 to 87] | 58.8 [27 to 88] | 59.7 [24 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 64 | 98
  Male | 67 | 131 | 198
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 101 | 195 | 296

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants (or Chart Reviews) With Complete Success of Primary Vitrectomy Surgery
Description: Complete success of primary vitrectomy surgery, defined as retinal re-attachment without the need for any additional surgical procedures.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab | Chart Review
Number analyzed (Participants) | 101 | 195
Participants | 92 | 169

2. Secondary Outcome: Number of Participants (or Chart Reviews) With Presence of Proliferative Vitreoretinopathy
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab | Chart Review
Number analyzed (Participants) | 101 | 195
Participants | 9 | 26

ADVERSE EVENTS:
Time Frame: up to 6 months
Description: Comparison arm is a retrospective cohort, no prospective intervention evaluated.
Arm/Group | Bevacizumab | Chart Review
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/0
Other Adverse Events (participants affected / at risk) | 0/101 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-18): https://cdn.clinicaltrials.gov/large-docs/70/NCT02192970/Prot_SAP_000.pdf